CLINICAL TRIAL: NCT04459221
Title: Study of the Impact of a School Program Combining - Promotion of HPV Vaccination and HPV Vaccine Offer in Middle School - on Adherence to HPV Vaccination in Middle School Students
Acronym: PROM SSCOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/CHU/05; 2020-002332-73 (EudraCT Number)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Papilloma Viral Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitating access to HPV vaccination (Experimental)
  Interventions: Drug: Gardasil 9, 9-Valent Intramuscular Suspension
- promotion of HPV vaccination (No Intervention)

INTERVENTIONS:
Drug: Gardasil 9, 9-Valent Intramuscular Suspension — access to HPV vaccination near the college in a health bus
  Arms: Facilitating access to HPV vaccination

SUMMARY:
Cervical cancer (CCU) is the fourth most common cancer in women worldwide. In Reunion island, CCU is the third leading cause of cancer in women (standardized incidence rate on the world population (TIS) in 2013 of 10.3 / 100,000) and is the eighth deadliest cancer with a rate standardized mortality of 4.8 / 100,000, almost three times higher than in mainland France where it was 1.7 / 100,000 in 2018.

CCU results from infection with the human papillomavirus (HPV), which is the most common sexually transmitted viral infection.

CCU prevention is mainly based on cervical smear screening and anti HPV vaccination (VHPV) which has demonstrated its effectiveness on the prevalence of HPV carriage, but also on incidence of condyloma or intermediate grade dysplasia. Since HPV is mainly transmitted sexually, it is important to vaccinate before the start of sex.

In Reunion island, the HPV vaccination coverage rate is the lowest in France, estimated by Public Health France at 8.1% among girls aged 16 years in 2018, while the already low national average was established 23.7%.

Thus, in view of the epidemiological situation in Reunion island (high incidence and mortality for the CCU, very low VHPV coverage rate), we thought it would be interesting to study the impact of a health promotion program sex and prevention of sexually transmitted infections (STIs) including papillomavirus-related pathologies, with a program to promote HPV vaccination among young students in middle school.

ELIGIBILITY:
Inclusion Criteria:

* schooled in one of the classes drawn at random in the 2 colleges selected for the study,
* members or beneficiaries of a social security scheme,
* having agreed to participate in the study and whose parents or holder (s) of parental authority have signed a free, informed and written consent.

Exclusion Criteria:

* under the age of 9, or over the age of 17 at inclusion,
* with hypersensitivity to the active substances or to any of the excipients of the vaccine (Gardasil 9®),
* with a permanent contraindication to vaccination.
* having already initiated the HPV vaccination (complete or incomplete scheme). Students with an incomplete vaccination schedule will be referred to their attending physician to complete the missing dose (s).
* pregnancy or breastfeeding (based on the declaration)

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change the vaccination rate in girls | 9 month
  Number of girls having completed a complete vaccination schedule. Hypothesis: the intervention under study should increase the rate of vaccinated

SECONDARY OUTCOMES:
increase the vaccination rate in all student | 9 month
  number of student having completed a complete vaccination schedule
increase the vaccination rate in all student | 9 month
  number of student having completed a incomplete vaccination schedule

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran PL, Chirpaz E, Boukerrou M, Bertolotti A. Impact of a Papillomavirus Vaccination Promotion Program in Middle School: Study Protocol for a Cluster Controlled Trial. JMIR Res Protoc. 2022 Jun 13;11(6):e35695. doi: 10.2196/35695. PMID 35700023